CLINICAL TRIAL: NCT04531020
Title: Incidence of Emergence Delirium in the PACU: Prospective Observational Trial
Brief Title: Incidence of Emergence Delirium in the PACU
Acronym: PACUDEL
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR FN Brno 2020/10
Record Dates: First submitted 2020-08-21; First posted 2020-08-28 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Emergence Delirium
Keywords: Emergence delirium; Anaesthesia; Paediatric patient
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at PACU: Patients undergoing elective surgical or diagnostic intervention admitted to PACU after postanaesthesia recovery
  Interventions: Diagnostic Test: PAED measurement

INTERVENTIONS:
Diagnostic Test: PAED measurement — The incidence of emergence delirium, defined as PAED score above 10 points minimally in one of the PAED score measurements. PAED score will be measured in 0., 5., 10., 15., and 20. minute after PACU admission.
  Other Names: PAED score measurement at PACU

SUMMARY:
Emergence delirium (ED) is serious complication in the postoperative period in paediatric anaesthesia, reported incidence is 20-60%. It is characterized by psychomotor and perception disorder with excitation of paediatric patients. Emergence delirium has impact on morbidity and even on mortality of paediatric patients in the postoperative period.

The potential risk factors for ED development include sevoflurane, which is the dominant anaesthetic agent used in the paediatric patients, and which is actually the only inhalation agent used for inhalation anaesthesia induction. The incidence of ED is higher in postoperative period, for example in the Post-anaesthesia Care Unit - PACU. Patients with ED are at higher risk of psychomotor anxiety, agitation, unintentional extraction of intravenous cannula, and nausea and vomiting. For the therapy of ED propofol, midazolam and eventually ketamine in a reduced dosage are used.

DETAILED DESCRIPTION:
After the approval of the study by the Ethics Committee of the University hospital Brno and registration of the protocol at clinicaltrials.gov, the incidence of emergence delirium (ED) using PAED, WATCHA and Richmond agitation and sedation scale (RASS) score in patients hospitalized in the post-anaesthesia care unit (PACU) after general anaesthesia, in the Departement of paediatric anaesthesia and intensive care unit, University Hospital Brno in the term from 1.9.2020 until 30.6.2021 will be measured.

Paediatric Emergence Delirium (PAED) score, WATCHA score and Richmond agitation and sedation scale (RASS) will be measured in 0., 5., 10., 15., and 20. minute after PACU admission and after obtaining RASS ≥ - 2 . Emergence delirium is defined as PAED score above 10 points. In the case of ED development, the duration of ED will be measured as well as the number of therapeutic interventions and the cumulative dose of administered sedatives. The average PAED, WATCHA, RASS scale will be reported, the incidence of postoperative nausea and vomiting (PONV) and the cumulative dose of administered antiemetics, the type of anaesthesia induction (inhalation vs. intravenous), type of anaesthesia (TIVA, combined, inhalational), length of the surgery, type of the surgery will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients after general anaesthesia hospitalized in the PACU in the term rom 1.9.2020 until 30.6.2021.

Exclusion Criteria:

* Patients in the age from 0 to 1 month.

Ages: 1 Month to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients after general anaesthesia hospitalized in the PACU
Sampling Method: Non-Probability Sample
Enrollment: 1421 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence delirium | up to 60 minutes after PACU admission
  The incidence of emergence delirium, defined as PAED score above 10 points and/or WATCHA score over 2 and or RASS over 1 minimally in one of the measurements. All measurements will be measured in 0., 5., 10., 15., and 20. minute after PACU admission. The first measurement (T0) will be intiated after first obtaining RASS over -2.

SECONDARY OUTCOMES:
The duration of ED | up to 60 minutes after PACU admission
  The cumulative duration of ED will be measured
The average PAED score | up to 60 minutes after PACU admission
  The average PAED score at PACU will be measured
The need for pharmacology intervention incidence | up to 60 minutes after PACU admission
  The need for pharmacology intervention - defined by the number of therapeutic interventions
incidence of postoperative nausea and vomiting (PONV) | up to 60 minutes after PACU admission
  incidence of postoperative nausea and vomiting (PONV) defined by the cumulative dose of administered antiemetics
type of anaesthesia induction (inhalation vs. intravenous) | up to 60 minutes after PACU admission
  type of anaesthesia induction (inhalation vs. intravenous) will be evaluated
type of anaesthesia (TIVA, combined, inhalational) | up to 60 minutes after PACU admission
  type of anaesthesia (TIVA, combined, inhalational) will be evaluated
length of the surgery | up to 60 minutes after PACU admission
  length of the surgery will be evaluated
type of the surgery | up to 60 minutes after PACU admission
  type of the surgery will be evaluated
cumulative dose of administered sedatives | up to 60 minutes after PACU admission
  the cumulative dose of administered sedatives
The average WATCHA score | up to 60 minutes after PACU admission
  The average WATCHA score at PACU will be measured
The average RASS score | up to 60 minutes after PACU admission
  The average RASS score at PACU will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, prof. MD., Ph.D., Study Chair — Faculty of medicince Masaryk University and University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: Undecided